CLINICAL TRIAL: NCT01614691
Title: Safety and Efficacy of SPARC1203 in Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLR_12_03
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- SPARC1203 low dose (Experimental)
  Interventions: Drug: SPARC1203
- SPARC1203 mid dose (Experimental)
  Interventions: Drug: SPARC1203
- SPARC1203 high dose (Experimental)
  Interventions: Drug: SPARC1203
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SPARC1203 — Active
  Arms: SPARC1203 high dose; SPARC1203 low dose; SPARC1203 mid dose
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study will assess safety and efficacy of SPARC1203 delivered via nasal spray in patients with allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 65 years (both inclusive) with history of seasonal allergic rhinitis and positive skin prick test

Exclusion Criteria:

* History or presence of perennial allergic rhinitis
* Upper or lower respiratory tract infection 2 weeks before Visit 2
* Significant pulmonary disease other than allergic rhinitis or mild asthma controlled by beta-2-agonists alone
* Immunizations or vaccinations within 4 weeks prior to Visit 1

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2012-06; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change in Total Nasal Symptom Score (TNSS) | Baseline and 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- SPARC Site 1, Hanover, Germany

REFERENCES:
- [Derived] Badorrek P, Hohlfeld JM, Krug N, Joshi A, Raut A. Efficacy and safety of a novel nasal steroid, S0597, in patients with seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2015 Oct;115(4):325-329.e1. doi: 10.1016/j.anai.2015.07.016. Epub 2015 Aug 11. PMID 26272281